CLINICAL TRIAL: NCT00728494
Title: Evaluation of Compliance of HCV Genotype 1 Infected Patients Receiving PegIntron / Rebetol in Conjunction With a Patient Assistance Program - Non Interventional Observational Study.
Brief Title: Compliance of HCV Genotype 1 Infected Patients Receiving PegIntron/Rebetol and a Patient Assistance Program (Study P04671)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04671
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Results first posted 2009-08-19 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin; Allied Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment and Patient Assistance Program: Patient assistance program was provided to the participants treated with PegIntron/Rebetol. The support program consisted of training by physicians or specialized nurses on the significance of treatment compliance, methods for managing adverse events, and correct drug administration, as well as informational materials and assistance in the management of adverse events.
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: Rebetol (ribavirin; SCH 18908); Behavioral: Patient Assistance Program
- Treatment Alone: PegIntron/Rebetol treatment only.
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: Rebetol (ribavirin; SCH 18908)

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b; SCH 54031) — Peginterferon alfa-2b will be administered according to the product's labeling.
  Other Names: PegIntron
Drug: Rebetol (ribavirin; SCH 18908) — Ribavirin will be administered according to the product's labeling.
  Other Names: Rebetol
Behavioral: Patient Assistance Program — The patient assistance program includes the following:
  * Training by physicians or specialized nurses.
  * Informational materials based on the "To beat HCV" program.
  * Management of specific side effects.
  Other Names: Support program
  Groups: Treatment and Patient Assistance Program

SUMMARY:
Enrolled patients will be recruited to two parallel groups during therapy for Hepatitis C. Patients in the first one will receive a patient assistance program, and patients in the second group will not. All patients will receive PegIntron and Rebetol according to label.

DETAILED DESCRIPTION:
Non-Probability Sample, Commercial product used according to EU label.

ELIGIBILITY:
Inclusion Criteria:

* According to PegIntron/Rebetol label.
* Only HCV genotype 1 infected patients will be enrolled in the study.

Exclusion Criteria:

* According to PegIntron/Rebetol label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic HCV.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment and Patient Assistance Program | Treatment Alone
Started | 60 | 39
Completed | 51 | 32
Not Completed | 9 | 7
Not completed — Adverse Event | 7 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lack of Efficacy | 2 | 4
Not completed — No data available | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment and Patient Assistance Program | Treatment Alone | Total
Number analyzed (Participants) | 60 | 39 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (12) | 42 (14) | 45 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 43
  Male | 35 | 21 | 56
Region of Enrollment [Number; unit: participants]
  Poland | 60 | 39 | 99

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Complete Treatment With PegIntron/Rebetol Therapy for Hepatitis C
Description: Participant adherence to therapy was compared between participants treated with PegIntron/Rebetol either with or without a patient assistance program
Time Frame: At the end of the 48-week treatment period
Measure: Number; unit: Participants
Arm/Group | Treatment and Patient Assistance Program | Treatment Alone
Number analyzed (Participants) | 60 | 39
Participants | 51 | 32

2. Secondary Outcome: Average Length of Treatment
Description: Participant adherence to therapy was compared between participants who received vs not received a patient assistance program in addition to their PegIntron/Rebetol treatment.
Time Frame: Maximum 48-week treatment duration
Measure: Number; unit: Participants
Arm/Group | Treatment and Patient Assistance Program | Treatment Alone
Number analyzed (Participants) | 60 | 39
Participants
  2-12 weeks | 6 | 5
  13-47 weeks | 3 | 2
  48 weeks and one of the drugs at a dose <80% | 13 | 9
  48 weeks and both drugs at a dose >=80% | 38 | 23

3. Secondary Outcome: Average Dosage of PegIntron
Description: Dosage of PegIntron was expressed in terms of micrograms of PegIntron received per kilogram of participant's body weight per week
Time Frame: Up to 48-week treatment duration
Measure: Mean (Standard Deviation); unit: micrograms/kg/week
Arm/Group | Treatment and Patient Assistance Program | Treatment Alone
Number analyzed (Participants) | 60 | 39
micrograms/kg/week | 1.46 (0.16) | 1.45 (0.25)

4. Secondary Outcome: Average Dosage of Rebetol
Description: Rebetol dosage was expressed in milligrams per kilogram of body weight per day.
Time Frame: Up to 48-week treatment duration
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Treatment and Patient Assistance Program | Treatment Alone
Number analyzed (Participants) | 60 | 39
mg/kg/day | 12.63 (1.72) | 12.01 (2.86)

5. Primary Outcome: The Number of Participants With a Sustained Virologic Response at 6 Months Post-treatment
Description: Sustained virologic response is defined as having an undetectable hepatitis C virus ribonucleic acid (HCV-RNA) at the end of treatment and 6 months post-treatment
Time Frame: Measured at 6 months post-treatment
Measure: Number; unit: Participants
Arm/Group | Treatment and Patient Assistance Program | Treatment Alone
Number analyzed (Participants) | 51 | 12
Participants | 29 | 7

6. Primary Outcome: The Number of Participants Who Relapsed at 6 Months Post-treatment
Description: Participants who relapse are defined as having an undetectable HCV-RNA at the end of treatment but detectable HCV-RNA at 6 months post-treatment
Time Frame: Measured at end of treatment and 6 months post-treatment
Measure: Number; unit: Participants
Arm/Group | Treatment and Patient Assistance Program | Treatment Alone
Number analyzed (Participants) | 51 | 12
Participants | 17 | 4

ADVERSE EVENTS:
Arm/Group | Treatment and Patient Assistance Program | Treatment Alone
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/39
Other Adverse Events (participants affected / at risk) | 39/60 | 28/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment and Patient Assistance Program (N=60) | Treatment Alone (N=39)
ANAEMIA (Blood and lymphatic system disorders) | 12 (15) | 10 (10)
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 3 (3)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2)
ASTHENIA (General disorders) | 4 (4) | 3 (3)
CHEST PAIN (General disorders) | 1 (1) | 3 (3)
FATIGUE (General disorders) | 4 (4) | 3 (3)
INFLUENZA LIKE ILLNESS (General disorders) | 6 (6) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 8 (11)
PNEUMONIA (Infections and infestations) | 0 (0) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 4 (5) | 0 (0)
WEIGHT DECREASED (Investigations) | 13 (14) | 7 (8)
APPETITE DISORDER (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 1 (1) | 2 (2)
DEPRESSION (Psychiatric disorders) | 5 (5) | 0 (0)
DYSTHYMIC DISORDER (Psychiatric disorders) | 0 (0) | 2 (3)
INSOMNIA (Psychiatric disorders) | 3 (3) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information obtained in the course of conducting the study, including all data concerning the study and its results, are confidential and cannot be disclosed to any third parties without the consent of Schering-Plough.